CLINICAL TRIAL: NCT02535962
Title: Effects of Probiotic Addition to Corticosteroid Treatment for PFAPA
Brief Title: Probiotics and Corticosteroids for Treating Periodic Fever, Aphthous Stomatitis, Pharyngitis, Cervical Adenitis (PFAPA)
Acronym: PFAPA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor withdrawal
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Principal Investigator, Nicholas Bennett, Medical Director of Infectious Disease Department, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-017
Record Dates: First submitted 2015-08-20; First posted 2015-08-31 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Periodic Fever; Aphthous Stomatitis; Pharyngitis; Cervical Adenitis
Keywords: PFAPA
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases; Stomatitis, Aphthous; Pharyngitis | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteriod + Probiotic Treatment (Experimental): Corticosteroid dosing of 1 mg/kg of body weight given once at the onset of the febrile period, repeated once within 24 hours if necessary, but no more than two doses per cycle. The second dose of corticosteroid treatment is only to be given within one day following the initial dosage if the fever persists.
  Investigational drug (Intervention is Lactobacillus acidophilus and Bifidobacterium lactis): Patients will be instructed to take one sachet of the study product mixed into a 60 ml of water that is not hot. Each sachet will contain Lactobacillus acidophilus NCFM and Bifidobacterium lactis Bi-07 at a dose of 5*109 CFU of each strain. The investigational product will be taken daily for the duration of the study, which is a year.
  Interventions: Biological: Lactobacillus acidophilus and Bifidobacterium lactis
- Corticosteriod + PlaceboTreatment (Placebo Comparator): Corticosteroid dosing of 1 mg/kg of body weight given once at the onset of the febrile period, repeated once within 24 hours if necessary, but no more than two doses per cycle. The second dose of corticosteroid treatment is only to be given within one day following the initial dosage if the fever persists.
  Placebo: will be taken daily and patients will be instructed to take one sachet of placebo mix into 60ml of water that is not to hot. The placebo will be taken daily for the duration of the study, which is one year. Placebo will be 1g of sucrose that has identical appearance, smell, and taste with the study product.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Lactobacillus acidophilus and Bifidobacterium lactis — study product will be freeze dried and put into foil sachets
  Other Names: HOWARU® Protect Kids
  Arms: Corticosteriod + Probiotic Treatment
Other: Placebo — Placebo will look and taste like the investigational product. This also will be provided in a foil sachets
  Arms: Corticosteriod + PlaceboTreatment

SUMMARY:
The purpose of study is to see if adding probiotics to corticosteroid treatment for children with PFAPA could improve the health and daily of patients through reduction in febrile period frequency and length, along with concomitant reduction of associated symptoms. Current standard of care incorporates the administration of corticosteroids; however, while limiting the symptoms associated with PFAPA, corticosteroid use has been shown to increase the frequency at which these symptoms occur. Investigators hypothesize that administration of probiotics along with corticosteroids will work to decrease the frequency at which the febrile episodes occur. Additionally, probiotics may decrease the maximal fever experienced during these episodes, amount of corticosteroid needed to control the symptoms, average length of the episodes, and the number of patients who ultimately undergo tonsillectomy due to unsuccessful treatment with medication.

DETAILED DESCRIPTION:
Periodic fever, aphthous stomatitis, pharyngitis, and cervical adenitis (PFAPA) was first described in 1987 in a study of 12 pediatric patients. PFAPA is predominately considered a pediatric illness with onset typically occurring under the age of 5. This syndrome is characterized by periodic febrile episodes (39°C - 42°C) lasting an average of 4 days with recurrence approximately every 21-30 days. Patients classically exhibit at least one of three major associated symptoms; aphthous stomatitis, pharyngitis, or cervical adenitis. Between periods of fever, patients are asymptomatic and do not experience long-term deleterious effects on growth or development. Currently, the etiology of this syndrome is unknown but does not appear to be heritable or target specific populations.

Due to a lack of applicable diagnostic tests, the identification of PFAPA is predominantly dependent on patient history and physical examination. This methodology relies heavily upon clinical presentation of the patient's illness to rule out other causes of periodic fever. As a result of the unknown cause of PFAPA, there are several proposed treatment approaches available. Corticosteroids are the current standard of care; typically a single dose of prednisolone (1 mg/kg), given upon first signs of fever with a subsequent dose during the febrile period if necessary. Several studies have shown that administration of prednisolone was sufficient to abort the febrile episode. However, this treatment method typically results in a decrease in the healthy interval between fever reoccurrence. The reduction in fever allows for children to attend school and participate in other activates, but the increased frequency provides additional complications for children and parents.

Oral cimetidine, a histamine H-2 receptor agonist that results in reduced production of stomach acid, has also been used as possible treatment. This treatment has shown to inhibit febrile episodes, it was only effective in <30% of patients.

If medication therapy fails to resolve recurrent febrile episodes, the option of tonsillectomy presents a possible alternative. PFAPA syndrome was shown to resolve in the majority of patients, however this not preferred as a first line treatment due to the risks associated with surgery and general anesthesia.

Recently published literature suggests a potential new treatment for PFAPA targeting chemokines and proinflammatory cytokines. A possible method for the inhibition of cyclic inflammatory responses in PFAPA would be the exposure of patients to a safe level of continuous low-grade inflammation, resulting from an immune response. In previous studies investigating allergy and eczema relief in pediatric populations, it was shown that administration of probiotics induced elevated levels of inflammatory markers. These low level inflammatory responses resulted in no adverse effects and provided an immunologic activation benefit. Use of probiotics provides a previously unstudied approach to the treatment of PFAPA. Dr. Nicholas Bennett has also observed anecdotal evidence that patients who self-administered probiotics experienced relief of their PFAPA symptoms.

This is a randomized, prospective, double-blind, placebo-controlled study with the randomization being done by the research pharmacist using an equal randomization process, no stratification of patients. Dr. Bennett and other patient recruiters will remain blinded to the participant group assignment. The standard of care consists of corticosteroid dosing of 1 mg/kg of body weight given once at the onset of the febrile period, repeated once within 24 hours if necessary, but no more than two doses per cycle. The second dose of corticosteroid is only to be given within one day following the initial dosage if the fever persists. The investigational product will be administered daily for the duration of the study. For the investigational product patients will be instructed to take daily one sachet of the study product mixed into a 60 ml of water that is not hot. On days 90±7, 180±7 and 270±7 patients will come to the study site for re-supply of the probiotic and for evaluation of compliance. Throughout the 1-year followup period, parents will be asked to keep a journal to track corticosteroid usage, probiotic usage, additional medication usage, fever intensity, and associated symptoms. Standardized thermometers will be provided to ensure consistency. These journals will be collected and patient progress will be monitored at the standard care visits every three months. In addition, follow-up phone calls will be made monthly to assess progress and to address any concerns.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis or confirmation of diagnosis of PFAPA from Dr. Bennett based on clinical or laboratory data
* is or will be undergoing treatment for PFAPA at CCMC
* agrees to the consent and, if necessary, assent forms
* is between 1 and 12 years of age

Exclusion Criteria:

* is currently taking another probiotic regularly (>=2 times/ week)
* is allergic to ingredients in the probiotic or placebo
* may react adversely to the probiotic due to any form of immune deficiency or chronic disease including pulmonary, renal, cardiac disorders including underlying structural heart disease, gastrointestinal disease, or diabetes
* is not a proficient English speaker
* does not agree to the consent and/or assent forms
* patients who use antibiotics or have used them within a month of the study start

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Effects of the investigational treatment | Time to event: number of fever-free days will be calculated, as well as the average number of days between fever cycles from baseline to end of study which is 12 months.
  Increased healthy intervals between cyclic febrile episodes in patients with PFAPA compared to patients being solely treated with corticosteroids.
Safety of the investigational treatment - reported descriptively as percentages of patients experiencing adverse and serious adverse events. | Time to event: number of fever-free days will be calculated, as well as the average number of days between fever cycles from baseline to end of study which is 12 months.
  Safety will be reported descriptively as percentages of patients experiencing adverse and serious adverse events.

SECONDARY OUTCOMES:
Maximal fever experienced during a PFAPA febrile episode will be recorded as an average of the peak temperature recorded during each episode throughout the year and compared between the study groups | Maximal fever experienced during a PFAPA febrile episode will be recorded as an average of the peak temperature recorded during each episode throughout the year
  Decreased maximal fever experienced during a PFAPA febrile episode.
Number of administrations of corticosteroid necessary for treatment of PFAPA syndrome, recorded as the average number of administrations per fever episode throughout the year | Number of administrations of corticosteroid necessary for treatment of PFAPA syndrome, recorded as the average number of administrations per fever episode throughout the year
  Decreased administrations of corticosteroid necessary for treatment of PFAPA syndrome.
The average duration of the individual cyclic febrile episodes | average duration of the individual cyclic febrile episodes in patients with PFAPA will be assessed from baseline to the end of study which is 1 year
  Decrease duration of the individual cyclic febrile episodes in patients with PFAPA.
The number of patients undergoing tonsillectomy will be compared between the study groups | At any time during the study from baseline to end of study, which is 12 months this will recorded
  Fewer patients undergoing tonsillectomy as a treatment for PFAPA syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bennett, MBBChir PhD, Principal Investigator — Connecticut Children's Medical Center